CLINICAL TRIAL: NCT06803927
Title: Non-Endoscopic Detection of Barrett's Esophagus and Esophageal Neoplasia Using Methylation Biomarkers on Endosign® Cell Collection Device Samples
Brief Title: Non-Endoscopic Detection of Barrett's Esophagus Using Methylation Biomarkers on EndoSign® Cell Collection Device Samples
Acronym: DETECT-ME
Status: Recruiting | Type: Observational
Sponsor: Cyted Health Inc (Industry)
Responsible Party: Sponsor
Other Study IDs: ENDOEXT-28
Record Dates: First submitted 2025-01-22; First posted 2025-01-31 (Actual); Last update posted 2025-08-21 (Actual); Status verified 2025-08

CONDITIONS: Barrett Esophagus
Keywords: Endosign® Cell Collection Device; Barretts Esophagus
MeSH Terms: conditions — Barrett Esophagus

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — DNA extracted from esophageal cells collected on the sponge.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- High Risk Screening without Barrett's Esophagus: Subjects with chronic GERD plus 3 other defined risk factors for Barrett's Esophagus (ACG) (e.g., age >50, male, white, obese, family history) who have had a standard of care endoscopy in which no Barrett's esophagus was identified.
  Interventions: Device: Barrett's Esophagus Test (LDT)
- Barrett's Esophagus: Subjects with known Barrett's esophagus with or without dysplasia/cancer identified or confirmed (surveillance) via a standard of care endoscopy
  Interventions: Device: Barrett's Esophagus Test (LDT)

INTERVENTIONS:
Device: Barrett's Esophagus Test (LDT) — Barrett's Esophagus Test (LDT) will be performed on esophageal cells collected using the EndoSign Cell Collection Device (510(k) cleared) and compared to the results of standard of care EGD plus biopsies (if applicable)

SUMMARY:
This study is looking at cells collected from the esophagus using a diagnostic device called the EndoSign® Cell Collection Device (a sponge on a thread). Subjects swallow a capsule, which dissolves in the stomach and releases a sponge that collects cells from the esophagus as the sponge is withdrawn using the thread. These cells will be tested to check for a condition called "Barrett's Esophagus."

The cells from the sponge will be tested using Cyted Health biomarkers and compared to the results from a regular endoscopy and any biopsies that are taken. To do this, we need sponge samples from people who might have Barrett's Esophagus based on their risk factors, and from people with Barrett's Esophagus.

Subjects will have one visit to have the Endosign Cell Collection Device administered prior to having a standard of care endoscopy. They will answer some questions about their medical history and experience with the cell collection procedure as part of the study. Data will be collected from medical records including post-endoscopy.

ELIGIBILITY:
High Risk Screening Inclusion Criteria

* Undergoing a standard of care EGD
* Willing to undergo non-endoscopic sampling with the study device prior to EGD (up to 6 weeks prior to EGD or same day as EGD).
* Willing and able to sign informed consent
* Must have chronic GERD as defined in the ACG Guidelines
* Must have at least 3 additional risk factors as defined in the ACG guidelines such as:
* Age ≥ 50
* Family history of Barrett's esophagus or esophageal adenocarcinoma
* Current or former smoker
* Obesity (BMI greater than or equal to 30 kg/m2)
* Male
* Non-Hispanic White

Exclusion Criteria

* Previous EGD for BE, with no BE identified
* Known BE or EAC
* Current dysphagia (unable to swallow a pill the size of the capsule (8.5 mm diameter))
* Known or suspected gastric or esophageal varices
* Known or suspected portal hypertension
* Taking anti-thrombotic medications that cannot be discontinued
* Taking GLP-1 agonists that cannot be discontinued for 1 week prior to sponge administration
* Previous gastric or esophageal surgery (including Nissen fundoplication)
* History of oropharyngeal tumor
* History of myocardial infarction or cerebrovascular accident in past 6 months
* Known or suspected to be pregnant (self-report for women of child-bearing potential)

Barrett's Esophagus Inclusion Criteria

* Undergoing a standard of care EGD (with or without endoscopic eradication therapy {EET})
* Willing to undergo non-endoscopic sampling with the study device prior to EGD (up to 6 weeks prior to EGD/EET or day of EGD/EET).
* Willing and able to sign informed consent
* Confirmed Barrett's Esophagus of length at least 1 cm or greater. This includes non-dysplastic Barrett's, low-grade dysplasia, high-grade dysplasia or adenocarcinoma.

Exclusion Criteria

* Previous EGD result was indefinite for dysplasia
* Previous endoscopic eradication therapy (EET)
* Current dysphagia (unable to swallow a pill the size of the capsule (8.5 mm dia.))
* Known or suspected gastric or esophageal varices
* Known or suspected portal hypertension
* Taking anti-thrombotic medications that cannot be discontinued
* Taking GLP-1 agonists that cannot be discontinued for 1 week prior to sponge administration
* Previous gastric or esophageal surgery (including Nissen fundoplication)
* History of oropharyngeal tumor
* History of myocardial infarction or cerebrovascular accident in past 6 months
* Known or suspected to be pregnant (self-report for woman of child-bearing potential)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects scheduled for EGD (upper endoscopy) that meet the eligibility criteria at recruiting centers.
Sampling Method: Non-Probability Sample
Enrollment: 700 (Estimated)
Dates: Start 2025-02-05 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Performance of Barrett's Esophagus Test (LDT) compared to standard of care. | Sample collection prior to standard of care endoscopy
  Performance of the biomarker for detecting BE or confirming no BE in the study population including sensitivity, specificity, negative predictive value (NPV), and positive predictive value (PPV) on samples collected using the EndoSign Cell collection device as compared to endoscopy and pathology.

SECONDARY OUTCOMES:
Assess subject experience with the EndoSign Cell Collection Device | Through the end of the study-about 9 months
  Use of a 10-point scale to assess subject's experience with the device where 0 is no issues and 10 is the worst experience on a number of device-specific questions

OTHER OUTCOMES:
Interim assessment of number of subjects with each diagnosis | Halfway through the study at about 4 months
  At 50% total recruitment to various diagnoses, the Sponsor will evaluate the number of subjects in that cohort with complete clinical data and sample collection. The Sponsor may issue notices to recruiting sites temporarily or permanently closing a cohort to new subjects.

CONTACTS AND LOCATIONS:
Overall Officials: Co-Lead Investigator, Principal Investigator — University of North Carolina; Co-Lead Investigator, Principal Investigator — University of Colorado, Denver
Locations (1):
- Gastroenterology Practice, Cordova, Tennessee, United States

IPD SHARING:
Plan to Share IPD: Undecided